CLINICAL TRIAL: NCT03804632
Title: A Prospective Observational Multi Center Study to Assess the Level of Asthma Control at Government Health Clinics (Klinik Kesihatan) in Malaysia.
Brief Title: Assessment of Asthma Control Level in Primary Care Setting in Malaysia
Acronym: ASCOPE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D2287R00120
Record Dates: First submitted 2019-01-14; First posted 2019-01-15 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Asthma Control Level

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GINA-defined clinical diagnosis of Asthma: All patients with GINA-defined clinical diagnosis of Asthma seen at respiratory clinic from October to December 2017 with age 18 and above

SUMMARY:
A prospective observational multi center study to assess the level of asthma control at Primary Care Setting; government health clinics (Klinik Kesihatan) in Malaysia. The specific objective of the study is to assess, in real-life clinical practice in Malaysia, the level of asthma control and the potential risk factors for uncontrolled disease in asthma patients treated at government health clinics.

DETAILED DESCRIPTION:
Despite the availability of GINA global guideline on asthma management which is widely referred by health care providers in Malaysia, the control of asthma is still a critical challenge. According to National Health and Morbidity Survey 2011, the prevalence of asthma in Malaysia is at 6.3%. Based on self-rated health status, 5.5% of patients were reported to be in good health whereas 9.9% reported poor health status although medications such as inhaled corticosteroids (ICS) and long-acting beta agonists (LABA) are widely available for effective asthma management. There is limited data to assess the level of asthma control at the Primary Care Setting in Malaysia which includes current clinical manifestation and future risk of exacerbation. Given the lack of data on Asthma control level, the awareness on the current disease control level will assist to properly characterise the patients based on GINA control level thus leading to appropriate diagnosis and treatment. The specific objective of the study is to assess, in real-life clinical practice in Malaysia, the level of GINA-defined asthma control and the potential risk factors for uncontrolled disease in asthma patients.

ELIGIBILITY:
Inclusion Criteria:

* Malaysians who have been diagnosed with Asthma by a physician verified by an investigator and seen at government health clinic (Klinik Kesihatan) from October - December 2017
* Be at least 18 years of age

Exclusion Criteria:

* Clinical features suggesting emphysema or chronic bronchitis and other chronic lung diagnosis
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatients seen and treated by health care providers at government health clinics.
Sampling Method: Non-Probability Sample
Enrollment: 1011 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-06-06 (Actual)

PRIMARY OUTCOMES:
Level of GINA-defined asthma control | up to 8 months
  GINA-defined asthma control: According to clinical characteristics that include daytime symptoms, limitations of activity, nocturnal symptoms/awakening, need for reliever/rescue treatment. Patient's are classified as controlled, partially controlled or uncontrolled.

SECONDARY OUTCOMES:
Types of medication prescribed for asthma control | up to 8 months
  Pharmacological management used for asthma control
Asthma control level | up to 8 months
  Asthma control is evaluated by patients' self-completion of the Asthma Control Test (ACT). The ACT is a reliable, valid tool that helps physicians identify patients with uncontrolled asthma in a clinical setting. The questionnaire assesses the frequency of asthma symptoms and patients' own perception of asthma control during the previous 4 weeks. Based on the sum of scores, complete asthma control (25 points), well-controlled asthma (20-24 points) or no asthma control (≤19 points) is revealed.
Adherence level in patients with inhalers | up to 8 months
  Adherence level measured by Malaysia Medication Adherence Scale (MALMAS)
  The first item of the MALMAS has five responses: (1) All the time, (2) Often, (3) Sometimes, (4) Rarely and (5) Never.
  The remaining seven items have a dichotomous response of "Yes" or "No". The responses in the MALMAS were scored based on the MMAS-8 where the total score ranged from 0 to 8. Both instruments categorized medication adherence based on the total scores obtained: low adherence (total score<6), medium adherence (6 to < 8) and high adherence (total score = 8)

CONTACTS AND LOCATIONS:
Locations (10):
- Malaysia (10):
  - Research Site, Port Dickson, Negeri Sembilan
  - Research Site, Seremban, Negeri Sembilan
  - Research Site, Pantai Remis, Perak
  - Research Site, George Town, Pulau Pinang
  - Research Site, Kota Kinabalu, Sabah
  - Research Site, Asajaya, Sarawak
  - Research Site, Banting, Selangor
  - Research Site, Rawang, Selangor
  - Research Site, Bandar Permaisuri, Terengganu
  - Research Site, Kuala Terengganu, Terengganu

REFERENCES:
- [Derived] Mohd Isa NA, Cheng CL, Nasir NH, Naidu V, Gopal VR, Alexander AK. Asthma control and asthma treatment adherence in primary care: results from the prospective, multicentre, non-interventional, observational cohort ASCOPE study in Malaysia. Med J Malaysia. 2020 Jul;75(4):331-337. PMID 32723990
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=14738&filename=ASCOPE_Synopsis_CTT.pdf